CLINICAL TRIAL: NCT02205606
Title: A Randomized, Double-Blind, Multicenter, Phase 3 Study to Evaluate Efficacy and Safety of HCP1306 Tablet in Patients With Primary Hypercholesterolemia
Brief Title: Efficacy/Safety of HCP1306 Tablet Versus HGP0816 Tablet in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ROZE-301
Record Dates: First submitted 2014-07-30; First posted 2014-07-31 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2014-07

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- HGP0816 5mg (Active Comparator)
  Interventions: Drug: HGP0816 5mg
- HGP0816 10mg (Active Comparator)
  Interventions: Drug: HGP0816 10mg
- HGP0816 20mg (Active Comparator)
  Interventions: Drug: HGP0816 20mg
- HCP1306 5/10mg (Experimental)
  Interventions: Drug: HCP1306 5/10mg
- HCP1306 10/10mg (Experimental)
  Interventions: Drug: HCP1306 10/10mg
- HCP1306 20/10mg (Experimental)
  Interventions: Drug: HCP1306 20/10mg

INTERVENTIONS:
Drug: HGP0816 5mg — P.O.
  Arms: HGP0816 5mg
Drug: HGP0816 10mg — P.O.
  Arms: HGP0816 10mg
Drug: HGP0816 20mg — P.O.
  Arms: HGP0816 20mg
Drug: HCP1306 5/10mg — P.O.
  Arms: HCP1306 5/10mg
Drug: HCP1306 10/10mg — P.O.
  Arms: HCP1306 10/10mg
Drug: HCP1306 20/10mg — P.O.
  Arms: HCP1306 20/10mg

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of HCP1306 in patients with primary hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 19 years
* Signed informed consent
* At visit 1, LDL-C ≤ 250mg/dL and Triglyceride < 400 mg/dL
* After 4 weeks more TLC, At visit2, LDL-C ≤ 250mg/dL, Triglyceride < 400 mg/dL and satisfied criteria according to Risk of cardiovascular disease

Exclusion Criteria:

* Current or past history of hypersensitivity to HMG-CoA reductase inhibitors and component of Ezetimibe
* Has an active liver disease and severe liver disorder (continous elevation of AST, ALT level or exceeds more than 3 times of normal upper limit)
* Has a severe renal failure and kidney injury (Creatinine level exceeds more than 2 times of normal upper limit)
* CK level exceeds more than 5 times of normal upper limit
* Uncontrolled hypertension patient (SBP≥ 180 mmHg or DBP ≥ 110 mmHg)
* Uncontrolled diabetes mellitus patient (HbA1c ≥ 9%)
* Uncontrolled malfunctional thyroidism (or at pre-visit 2, TSH level exceeds more than 1.5 times of normal upper limit)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline to 8 week in LDL-Cholesterol | baseline and 8 week

SECONDARY OUTCOMES:
Percent change from baseline to 4 week in LDL-Cholesterol | baseline and 4 week
Percentage of patients reaching treatment goals according to NCEP ATP III Guideline | week 4, week 8
Percent change from baseline to 4 week and 8 week in TC | week 4, week 8
Percent change from baseline to 4 week and 8 week in HDL-C | week 4, week 8
Percent change from baseline to 4 week and 8 week in TG | week 4, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-soo Kim, MD, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- 19 institutions including Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Rhee MY, Kim KJ, Kim SH, Yoon YW, Rha SW, Hong SJ, Kwak CH, Kim W, Nam CW, Park TH, Hong TJ, Park S, Ahn Y, Lee N, Jeon HK, Jeon DW, Han KR, Moon KW, Chae IH, Kim HY, Kim HS. Ezetimibe and Rosuvastatin Combination Treatment Can Reduce the Dose of Rosuvastatin Without Compromising Its Lipid-lowering Efficacy. Clin Ther. 2019 Dec;41(12):2571-2592. doi: 10.1016/j.clinthera.2019.10.010. Epub 2019 Nov 11. PMID 31727361